CLINICAL TRIAL: NCT06922786
Title: Hemadsorption to Enhance Drug Elimination in Intoxications
Acronym: MATRIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Michaël Mekeirele, Medical Doctor, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-24-12-050174
Record Dates: First submitted 2025-04-02; First posted 2025-04-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Intoxication by Drug
Keywords: Benzodiazepine; Tricyclic antidepressant; Intoxication; Hemadsorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hemadsorption (Experimental): Hemadsorption via a dialysis catheter will be performed in patients who are unconscious due to an intoxication with quantifiable benzodiazepines or tricyclic antidepressants 8 hours after admission. Before and after application fo this hemadsorption filter plasma titers of this drug will be obtained. After application of the hemadsorption filter pre- and post-filter titers will be obtained.
  Interventions: Device: Hemadsorption filter

INTERVENTIONS:
Device: Hemadsorption filter — Plasma titers neurodepressing drug:
  * At admission to the hospital (standard of care)
  * 2 hours after admission (+/- 15 minutes)
  * 4 hours after admission (+/- 15 minutes)
  * 6 hours after admission (+/- 15 minutes)
  * 8 hours after admission (+/- 15 minutes)
  * Just before start hemadsorption
  Hemadsorption via dialysis catheter in patients still fulfilling inclusion criteria 8 hours after admission.
  Subsequent plasma titers pre- and post-hemadosorption filter:
  * 15 minutes after start of hemadsorption (+ 15 minutes)
  * 4 hours after start of hemadsorption (+/- 15 minutes)
  * 8 hours after start of hemadsorption (+/- 15 minutes)
  * 12 hours after start of hemadsorption (+/- 15 minutes)
  * 16 hours after start of hemadsorption (+/- 15 minutes)
  * 20 hours after start of hemadsorption (+/- 15 minutes)
  * 24 hours after start of hemadsorption (+/- 15 minutes)
  * Every other 24 hours until cessation of hemadsorption or normalization of the plasma titer (+/- 15 minutes)

SUMMARY:
In this trial the investigators assess the effectiveness of applying a hemadsorber (cytosorb®) in removing benzodiazepines or tricyclic antidepressants in intoxicated patients admitted to ICU with prolonged impaired consciousness. This is a one arm interventional investigation where a hemadsorption filter is applied in patients fulfilling inclusion criteria 8 hours after admission. Plasma titer of the neurodepressing drug will be collected sequentially both before and after start of hemadsorption to evaluate the speed of drug elimination before and after application of a hemadsorption filter. Pre- and post filter titers will be obtained to evaluate adsorbability and to evaluate time to saturation of the filter.

DETAILED DESCRIPTION:
In this prospective interventional study with medical device, the investigotors would include 18 patients admitted to ICU after an intoxication with a quantifiable neurodepressing drugs (type benzodiazepines or tricyclic antidepressants) and with impaired consciousness defined as need for intubation or need for Flumazenil to prevent intubation. Naloxone is administered per standard of care to identify if opioid intoxications is the main reason of neurodepression. Patients requiring mechanical ventilation for other reasons than impaired consciousness due to this intoxication or indication for prolonged use of sedatives are excluded.

Patients with at least one risk factor for delayed drug elimination (Chronic kidney disease G3b or CHILD-Pugh B or C) and persisting impaired consciousness after eight hours (including patients with persisting need for flumazenil) and having 5 plasma titers of the neurodepressing drug with intervals of 2 hours will be initiated on a hemadsorption filter after contact between the treating team and either dr. Michaël Mekeirele or dr. Tim Balthazar to verify inclusion criteria. Patients fulfilling inclusion criteria but lacking the 5 plasma titers will get additional plasma titers with intervals of 2 hours until 5 plasma titers are obtained. If these patients still fulfill inclusion criteria at that time then a hemadosorption filter will be initiated.

After starting hemadsorption a plasma titer pre- and post filter will be obtained after 15 minutes and every 4 hours after starting hemadsorption for the first 24 hours. After this timepoint additional plasma titers will be obtained every 24 hours until stopping hemadsorption or normalisation of the plasma titer.

ELIGIBILITY:
Inclusion Criteria:

1. older than18 years
2. Admission to ICU
3. GCS < 8 or requiring Flumazenil 8 hours after hospital admission
4. Having an intoxication with a benzodiazepine or tricyclic antidepressant that we can measure/quantify
5. Having a risk factor for delayed drug elimination defined as either Cirrhosis CHILD B/C or chronic kidney insufficiency KDIGO 3b or worse

Exclusion Criteria:

1. Pregnant patient
2. Patients in chronic dialysis before admission
3. Need for mechanical ventilation for other reasons than intoxications (e.g. pneumonia, neurotrauma)
4. Concomitant pathology requiring continued intravenous sedation
5. Known history of seizures
6. Contra-indication to heparin use
7. DNR restricting the use of mechanical ventilation or dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Difference in time to upper limit of normal of the dosed drug with versus without hemadsorption | From enrollment to the end of treatment (cesation hemadsorption) +/- 3 days
  Based on plasma titers before start of hemadsorption the half life of the drug can be calculated. A theoretical intersection with the upper boundary of normal of the intoxicated drug plasma titer can be calculated. This will be statistically compared to the real time of attaining this titer after start of hemadsorption.

SECONDARY OUTCOMES:
Adsorbability of the individual neurodepressing drugs | From enrollment to the end of treatment (cesation hemadsorption) +/- 3 days
  Comparing the pre- and post filter titer of the neurodepressing drug the adsorbability can be observed.
Time to saturation of hemadsorption filter | From enrollment to the end of treatment (cesation hemadsorption) +/- 3 days
  Comparing the pre- and post filter titer of the neurodepressing drug the time to saturation can be observed
Catheter related complications | From enrollment to the removal of the dialysis catheter +/- 3 days
  Catheter related complications (eg bleeding, infection) will be noted
Seizures during hemadsorption therapy | From enrollment to the end of treatment (cesation hemadsorption) +/- 3 days
  Seizures during hemadsorption therapy will be noted
Bleeding during hemadsorption therapy | From enrollment to the end of treatment (cesation hemadsorption) +/- 3 days
  Bleeding during hemadsorption therapy will be noted
Cost effectiveness of applying a Cytosorb® hemadsorption filter | From enrollment to discharge from ICU (+/- 1 week)
  Duration of ICU stay, duration of ventilation, cost of a hemadsorption filter and disposables amongst others will be used for an evaluation of cost effectiveness
Duration mechanical ventilation | From enrollment to extubation (+/- 3 days)
  Time to extubation and stop of flumazenil will be noted
Duration ICU stay | From enrollment to discharge from ICU (+/- 1 week)
  Time to discharge will be noted
Need and duration vasopressors | From enrollment to stop of vasopressors (+/- 3 days)
  Time untill discontinuation of vasopressors will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Michaël Mekeirele, Medical Doctor, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
Single center study